CLINICAL TRIAL: NCT04432506
Title: Pilot Study of Anakinra to Mitigate CAR-T Toxicity in Subjects With Relapsed or Refractory Large B-Cell Lymphoma
Brief Title: Anakinra for the Reduction of CAR-T Toxicity in Patients With Relapsed or Refractory Large B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1051; NCI-2020-04369 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1051 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent High Grade B-Cell Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, Large B-Cell, Diffuse | interventions — Interleukin 1 Receptor Antagonist Protein; Receptors, Interleukin-6; axicabtagene ciloleucel; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cyclophosphamide, fludarabine, axi-cel, anakinra) (Experimental): Patients receive cyclophosphamide IV over 60 minutes and fludarabine IV over 30 minutes on days -5 to -3 in the absence of disease progression or unacceptable toxicity. Patients then receive axicabtagene ciloleucel IV over 30 minutes or less on day 0 and anakinra SC on days 0-6 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anakinra; Biological: Axicabtagene Ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Anakinra — Given SC
  Other Names: Kinaret; Kineret; rIL-1ra; rIL1RN
Biological: Axicabtagene Ciloleucel — Given IV
  Other Names: KTE C19; KTE-C19; KTE-C19 CAR; Yescarta
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa

SUMMARY:
This phase II trial studies the side effects and best dose of anakinra and to see how well it works in reducing side effects (toxicity) associated with a CAR-T cell treatment called axicabtagene ciloleucel in patients with large B-cell lymphoma that has come back (relapsed) or has not responded to treatment (refractory). Anakinra is a drug typically used to treat rheumatoid arthritis but may also help in reducing CAR-T cell therapy toxicity. Giving anakinra in combination with axicabtagene ciloleucel may help control relapsed or refractory large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess safety and tolerability of anakinra in reducing incidence of cytokine release syndrome (CRS) within 30 days after infusion of chimeric antigen receptor (CAR) T cells in subjects with relapsed or refractory large B-cell lymphoma.

SECONDARY OBJECTIVES:

I. To determine incidence of all grades and duration of both CRS and immune-cell associated neurotoxicity syndrome (ICANS).

II. To determine the complete response rate (CRR), overall response rate (ORR), progression-free survival (PFS) and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To determine the effects of anakinra on the cytokine and chemokine profile in peripheral blood after CAR-T therapy.

II. To determine the effects of anakinra on the expansion and persistence of CAR T cells.

III. To correlate baseline characteristics with toxicity, response and survival after anakinra combined with CAR-T therapy.

OUTLINE: This is a dose-escalation study of anakinra.

Patients receive cyclophosphamide intravenously (IV) over 60 minutes and fludarabine IV over 30 minutes on days -5 to -3 in the absence of disease progression or unacceptable toxicity. Patients then receive axicabtagene ciloleucel IV over 30 minutes or less on day 0 and anakinra subcutaneously (SC) on days 0-6 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 and 4 weeks, and then at 2, 3, 6, 9, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory diffuse large B-cell lymphoma (DLBCL), primary mediastinal B-cell lymphoma (PMBCL), transformed follicular lymphoma (tFL), or high-grade B-cell lymphoma (HGBCL), at least 2 prior lines of systemic therapy
* Planned to receive standard of care therapy with axicabtagene ciloleucel
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease of >= 1.5 cm
* At least two weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for axicabtagene ciloleucel (axi-cel) therapy, except for systemic immune checkpoint inhibitory / immune stimulatory therapy. At least 3 half-lives must have elapsed from any prior systemic immune checkpoint inhibitory / immune stimulatory therapy at the time the subject is planned for leukapheresis (e.g. ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists, etc)
* Toxicities due to prior therapy must be stable and recovered to =< grade 1 (except for clinically non-significant toxicities such as alopecia)
* Absolute neutrophil count of >= 1.0 x 10^9/L
* Platelet count of >= 60 x 10^9/L
* Creatinine clearance (as estimated by Cockcroft Gault) >= 45 mL/minute (min)
* Serum alanine transaminase (ALT) / aspartate transaminase (AST) =< 2.5 upper limit of normal (ULN)
* Total bilirubin =< 1.5 mg/dL, except in subjects with Gilbert's syndrome
* Cardiac ejection fraction >= 50% with no evidence of pericardial effusion
* Baseline oxygen saturation > 92% on room air
* No evidence, suspicion, and/or history of lymphoma involving the central nervous system (CNS)
* Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)

Exclusion Criteria:

* History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 3 years
* History of Richter's transformation of chronic lymphocytic leukemia (CLL)
* Autologous stem cell transplantation within 6 weeks of planned axi-cel infusion
* History of allogeneic stem cell transplantation
* Prior CD19 targeted therapy
* Prior chimeric antigen receptor therapy or other genetically modified T cell therapy
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management. Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the principal investigator
* Known history of infection with human immunodeficiency virus (HIV) or hepatitis B (hepatitis B virus surface antigen [HBsAg] positive) or hepatitis C virus (anti-HCV positive). A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing
* Known history of tuberculosis. A negative Quantiferon or purified protein derivative (PPD) up to 2 months before start of anakinra is enough if no specific risk factors
* Presence of any indwelling line or drain (e.g., percutaneous nephrostomy tube, indwelling foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter). Dedicated central venous access catheters such as a Port-a-Cath or Hickman catheter are permitted
* Subjects with detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of CNS lymphoma, cerebrospinal fluid malignant cells or brain metastases
* History or presence of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
* Subjects with cardiac atrial or cardiac ventricular lymphoma involvement
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment
* Requirement for urgent therapy due to tumor mass effects such as bowel obstruction or blood vessel compression
* Primary immunodeficiency
* History of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment
* Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
* History of severe immediate hypersensitivity reaction to any of the agents used in this study, including E coli-derived proteins
* Live vaccine =< 6 weeks prior to planned start of conditioning regimen
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant
* Subjects of both genders who are not willing to practice birth control from the time of consent through 6 months after the completion of anakinra injections
* In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation Trial Treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Strati, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Anakinra Dose Level 1 (100 mg SQ daily x 7 days starting on Day 0)
- Cohort 2: Anakinra Dose Level 2 (100 mg SQ BID x 7 days starting on Day 0)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 6 | 10 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Any Grade Cytokine Release Syndrome (CRS)
Description: Will be tabulated according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version (v)5.0. CRS will be assessed by both Lee 2014 criteria as well as American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading system.
Time Frame: Within 30 days after infusion of CAR T cells
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 10 | 10
Participants | 10 | 9

2. Secondary Outcome: Incidence of Different Grades and Duration of Both CRS and Immune Cell-associated Neurotoxicity Syndrome (ICANS)
Description: Will be tabulated according to the NCI CTCAE v5.0. CRS will be assessed by both Lee 2014 criteria as well as ASTCT Consensus Grading system. ICANS will be assessed by both CTCAE v5.0 as well as ASTCT Consensus Grading system.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 10 | 10
Participants
  CRS | 10 | 9
  ICANS | 4 | 3

3. Secondary Outcome: Overall Response Rate
Description: Will be assessed using the Cheson 2014 Lugano Classification response criteria for malignant lymphoma.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 10 | 10
Participants | 8 | 9

4. Secondary Outcome: Complete Response Rate
Description: Will be assessed using the Cheson 2014 Lugano Classification response criteria for malignant lymphoma.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 10 | 10
Participants | 8 | 5

5. Secondary Outcome: Progression Free Survival
Description: Will be assessed using the Cheson 2014 Lugano Classification response criteria for malignant lymphoma. Will be estimated using the method of Kaplan and Meier.
Time Frame: From the start of treatment to disease progression or death due to any cause whichever happened first, assessed up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 10 | 10
Participants | 5 | 6

6. Secondary Outcome: Overall Survival
Description: as for outcome 5
Time Frame: From the start of treatment to death due to any cause, assessed up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 10 | 10
Participants | 5 | 8

ADVERSE EVENTS:
Time Frame: up to 24 months
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 5/10 | 2/10
Serious Adverse Events (participants affected / at risk) | 6/10 | 4/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=10)
Encephalopathy (Nervous system disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (General disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=10)
Neutropenia (Investigations) | 6 (6) | 8 (8)
Thrombocytopenia (Investigations) | 6 (6) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 10 (11)
Infections (Infections and infestations) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Hypotension (Vascular disorders) | 6 (6) | 1 (1)
Hypofibrinogenemia (Investigations) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 9 (9) | 7 (7)
Nausea (Gastrointestinal disorders) | 5 (5) | 8 (8)
Fatigue (General disorders) | 5 (5) | 8 (8)
Headache (Nervous system disorders) | 5 (5) | 6 (6)
Pain (General disorders) | 3 (3) | 6 (6)
Sinus Tachycardia (Cardiac disorders) | 4 (4) | 3 (3)
ALT increased (Investigations) | 3 (3) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
AST increased (Investigations) | 3 (3) | 1 (1)
Arrhythmia (Cardiac disorders) | 3 (3) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Insomnia (Nervous system disorders) | 2 (2) | 2 (2)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Serosal effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 1 (1) | 2 (2)
Tremors (Nervous system disorders) | 2 (2) | 1 (1)
CMV infection (Infections and infestations) | 2 (2) | 0 (0)
Bilirubin increased (Investigations) | 1 (1) | 0 (0)
Agitation (Nervous system disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04432506/Prot_SAP_000.pdf